| | Increasing the winter community participation of older adult wheelchair users | 1 |
|---|---|---|
| Increasing the winter community | participation of older adult wheelchair users | |
| NCT02622828 | | |

Increasing the winter community participation of older adult wheelchair users

Participation has been defined by the World Health Organization as "involvement in a life situation" and includes involvement in community, social, and civic realms. The concept of participation is more complex that simply considering the extent to one does or does not engage in a prescribed activity, rather it also has qualitative attributes that relate to the nature and self-perceived meaning of participation.<sup>2</sup> Research has supported the association between community participation among people with disabilities, and outcomes such as higher subjective ratings of quality of life and independence, improved sense of belonging, and positive self-perception of health.<sup>3-5</sup>

In Canada, 1.2 million people use mobility aids, such as wheelchairs, as a means to participate and engage in meaningful occupations within their community. Furthermore, the prevalence of mobility issues reported increases as people age, with approximately one-quarter of Manitobans age 75 or over reporting mobility issues. However, users of wheeled mobility devices (WMD) face numerous environmental barriers to community participation including barriers such as limited access to accessible public transportation, 8 lack of or poorly maintained ramps, 8-11 lack of accessible parking, 8 negative societal attitudes.<sup>8</sup> and lack of enforcement of accessibility regulations.<sup>12</sup>

One environmental barrier that WMD users in Manitoba acutely experience is winter weather. In a web-based survey of 99 Manitoban WMD users, <sup>13</sup> 80% of respondents reported needing additional help for home maintenance, transportation, and community access in the winter; however 57% reported not receiving that needed help. Respondents reported that limited community participation in winter led to feelings of loneliness, isolation, fear, and anxiety. Forty-two percent of respondents reported reducing their community participation frequency from almost daily in summer, to once or twice a week (or less) in winter; this finding was associated with older adult WMD users and those who lack access to family/friends for transportation. These results are particularly concerning, given a recent systematic review of community-dwelling older adults that provides strong evidence to support the positive impact of involvement in social, recreational, spiritual, and physical activity on health and quality of life.<sup>14</sup>

Though we are beginning to gain an understanding of participation barriers specific to WMD users in the winter, few studies have sought to address these barriers through the development of new technology or adapting environmental features. 15-17 The five environmental domains identified by International Classification of Functioning, Health and Disability (ICF)<sup>18</sup> (i.e., technological, natural, physical, social/attitudinal, and policy) interact with a person with a health condition to either promote or limit activity and participation. Targeted interventions directed toward one or more of those domains may be an effective way of addressing reduced winter community participation. The purpose of this study is to examine whether intervention strategies targeted at the level of the environment can successfully promote the community participation experiences of community-dwelling older adult *Manitobans who use WMD in the winter.* The findings of this pilot study will help determine the feasibility of, and guide the development of, a proposal targeted at conducting a larger scale study.

## **Method**

Overview Using a single-subject design, five older adult WMD users will each select three communitybased participation goals to work on throughout the winter months. Each participant will work with an occupational therapist to receive individually-focused interventions aimed at increasing community participation. A client-centred outcome measure will be used to set initial goals, and to measure change in performance and satisfaction with performance.

**Detailed Description** Given the subjective nature of participation the experience of participating, community-based interventions should consider the individual nature of participation occupations and strive to engage individuals in occupations considered meaningful to them. <sup>14</sup> This study will use an Interrupted Time Series Design (ITS), a quasi-experimental single-subject design suitable for evaluating the effectiveness of individually-designed interventions. 19 Using ITS, each participant serves as his/her

own control, multiple baseline measurements are taken, and multiple measures of the targeted outcome are collected throughout the study trajectory.<sup>20</sup>

# **Participants**

This application is a pilot study, and thus feasibility of the research approach will be examined by recruiting five older adult Manitobans who are wheelchair users. Participants will be recruited through collaboration with one or more of the five Winnipeg Regional Health Authority ACCESS Centres and other health resource centres for seniors including Active Living Coalition for Older Adults (ALCOA), Age and Opportunity, Creative Retirement Manitoba, Healthy Aging Resource Team (HART) and the Independent Living Resource Centre (ILRC). Posters will be used to recruit participants. Participants will be screened for inclusion by the occupational therapist using the Geriatric Depression Scale-Short Form<sup>21</sup> (GDS-SF) and the Montreal Cognitive Assessment<sup>22</sup> (MOCA). Inclusion criteria include: age 70 or older, user of a manual or power wheelchair or scooter for outdoor mobility, self-identifies a reduction in community participation throughout the winter months, community-dwelling, GDS-SF score of 5 or less, MOCA score >26, and lives within the perimeter of Winnipeg. If the score on the GDS-SF is >5 (indicating mild depression), the individual will not be included in the study and with permission of the individual, the occupational therapist will telephone the individual's physician and suggest further assessment.

#### **Measures**

The Canadian Occupational Performance Measure 23 (COPM) is a client-centered outcome measure designed to detect changes in performance and satisfaction in occupations that the individual has selfidentified as being important and difficult to perform. The COPM has well-established psychometric properties and will be used as the primary outcome measure and will be used to set treatment goals, determine baseline stability, and detect change in performance of, and satisfaction with, the goals. The Activity Card Sort <sup>24</sup>(ACS) uses a Q-sort methodology where photographs of people performing various activities are sorted into categories that the participant indicates interest in performing. The ACS will be used to identify valued instrumental, leisure and social activities that the person has performed in the past and/or desires to participate in in the future and will guide the formation of goals on the COPM. The WHO-DAS 2.0<sup>25</sup> is a generic self-report health status measure, linked to the concepts of health and disability outlined in the ICF and intended to identify limitations in six domains, including self-care, and community and social functioning experienced over the past 30 days. The WHO-DAS 2.0 is responsive to change, has excellent internal consistency, established content validity, and high convergent validity. The WHO-DAS 2.0 will be used to identify changes in overall health status that occur through the study. Follow-up semi-structured interviews will be conducted at the end of the intervention phase, to gain the perspective of each participant of the experience and personal value of working to increase winter community participation. Interview questions will address barriers and supports to participating in selfidentified occupations and impact on sense of inclusion and engagement in the community.

Procedure (repeated for each of 5 participants, entered concurrently into study)

| Recruit/screen for inclusion | Week 0 | Occupational therapist will conduct |
|---|---|---|
| ACS; COPM goal-setting phase | | initial assessment to establish goals |
| WHO-DAS 2.0 | | using the ACS and COPM. |
| COPM baseline measurements | Weeks 1-4 | Minimum 24 data points required to |
| (2x/week) | | conduct statistical analysis <sup>19</sup> |
| Intervention related to goal 1 (e.g. attend | Weeks 5-7 | A sample intervention for goal 3 |
| weekly spiritual services at local place | | might include working with |
| of worship) | | participant to: identify appropriate |
| Continue with baseline measurements | | neighborhood grocery store suitable |
| (2x/week) for goals 2 and 3 | | for mobility/accessibility needs (e.g. |

| Intervention for goal 2 (e.g. participate | Weeks 8-10 | store that has scooter and basket |
|---|---|---|
| in wheelchair yoga class 1x/week) | | available for customer use), |
| Continue with baseline measurements | | determine regular transportation |
| (2x/week) for goal 3 | | means and travel route, prepare |
| Intervention for goal 3 (e.g. weekly | Weeks 11-13 | weekly grocery list, learn to use debit |
| grocery shopping at local grocery store) | | card to pay for groceries. |
| Follow up phase (COPM/WHO-DAS) | Weeks 16 | Research assistant conducts follow up |
| Follow-up interview (week 16 only) | and week 20 | interviews and administer follow-up |
| | | COPM and WHO-DAS 2.0 |

# **Analysis**

COPM data will be plotted and visually inspected to gain an understanding of the timing and nature of any change. Statistical analysis will be conducted using the celeration line and C statistic 19, where the proportion of data points above and below the line is calculated and compared to a probability table to determine statistical significance. Repeated measures ANOVA will be used to identify change on the six domains of the WHO-DAS 2.0. Guided by an Interpretive Descriptive approach<sup>26</sup>, qualitative interviews will be transcribed verbatim and directed content analysis<sup>27</sup> used to gain a descriptive and interpretive understanding of clinically relevant issues and suggestions for future study.

# **Importance and Relevance to Aging**

Approximately one-third of Manitobans aged 65 or over reported emotional and social loneliness and older adults reported a decline in leisure activity participation with increasing age. Older adult WMD users in Manitoba bear a disproportionate burden in the winter – when aging, mobility limitations, and weather coincide to create conditions not conducive to community participation. A recent systematic review identified strong evidence to support the use of occupation and client-centred interventions in maintaining instrumental activities of daily living abilities of community-dwelling older adults.<sup>28</sup> However, evidence is required to identify whether, and how, we can use individually-focused interventions at the level of the environment to improve or maintain the community participation experiences of community-dwelling older adults who use WMD, <sup>28</sup> particularly in the winter.

# **Qualifications and Strategic New Direction**

My program of research focuses on understanding the intersection between assistive technology users and their environments. I primarily use client-centered approaches to inquiry, specifically qualitative methods, photovoice, case study, and mixed methods. While aging has not been a particular focus in past research, findings from a recent survey that I conducted<sup>13</sup> indicated a disproportionate burden placed on older adults who are WMD users in terms of limitations in community participation in winter. I view this application as an important opportunity to explore innovative ways of addressing those challenges.

## **Publications and Future Applications**

One peer-reviewed publication and a minimum of two professional presentations on this research will result from this study. While the sample size of five will not provide evidence of a treatment effect, the findings can be used to determine sample size required for a larger scale study proposal targeted at the Canadian Institutes of Health Research. This study will form a key component of a larger program of research focused on improving winter community participation among people with disabilities.

## **Timeline**

| Hire research assistant and OT; Submit HREB | July –August 2015 |
|---------------------------------------------|--------------------------|
| Recruit/Baseline phase | November – December 2015 |
| Intervention (to occur over mid-winter) | January - March 2016 |
| Follow up | Complete by April 2016 |

| Data analysis | Complete by July 2016 |
|----------------------------|-----------------------|
| Presentations/publications | May –September 2016 |

## References

- 1. World Health Organization. International Classification of Functioning, Disability, and Health 2001 [cited 2014 Apr 15]. Available from: URL: http://apps.who.int/classifications/icfbrowser/.
- 2. Law, M. (2002). Participation in the occupations of everyday life. American Journal of Occupational *Therapy*, 56(6), 640-649
- 3. Dattilo, J., Estrella, G., Estrella, L. J., Light, J., McNaughton, D., & Seabury, M. (2008). "I have chosen to live life abundantly": Perceptions of leisure by adults who use augmentative and alternative communication. Augmentative and Alternative Communication, 24(1), 16-28.
- 4. Levasseur, M., Desrosiers, J., & Noreau, L. (2004). Is social participation associated with quality of life of older adults with physical disabilities? Disability & Rehabilitation, 26(20), 1206-1213.
- 5. Milner, P., & Kelly, B. (2009). Community participation and inclusion: people with disabilities defining their place. Disability & Society, 24(1), 47-62.
- 6. Prevalence of Disability in Canada 2006: Analytical Report. Ottawa (ON); Statistics Canada. 2008. Catalogue No. 89-682-XWE- No.2.
- 7. Centre on Aging (2010). Profile of Manitoba's Seniors. Author: Winnipeg, MB
- 8. Wee, J., & Paterson, M. (2009). Exploring how factors impact the activities and participation of persons with disability: Constructing a model through grounded theory. The Qualitative Report, *14*(1), 165-200.
- 9. Brandt, A., Iwarsson, S., & Stahle, A. (2004). Older people's use of powered wheelchairs for activity and participation. Journal of rehabilitation medicine, 36(2), 70-77.
- 10. Chaves, E. S., Boninger, M. L., Cooper, R., Fitzgerald, S. G., Gray, D. B., & Cooper, R. A. (2004). Assessing the influence of wheelchair technology on perception of participation in spinal cord injury. *Archives of physical medicine and rehabilitation*, 85(11), 1854-1858.
- 11. Barker, D. J., Reid, D., & Cott, C. (2006). The experience of senior stroke survivors: factors in community participation among wheelchair users. Can J of Occupational Therapy, 73(1), 18-25.
- 12. Hammel, J., Jones, R., Gossett, A., & Morgan, E. (2006). Examining barriers and supports to community living and participation after a stroke from a participatory action research approach. *Topics in Stroke Rehabilitation*, 13(3), 43-58.
- 13. Ripat, J., Brown, C., & Ethans, K. Barriers to wheelchair use in the winter. Manuscript submitted for publication.
- 14. Stay, W. B., Hallenen, T., Lane, J., & Arbesman, M. (2012). Systematic review of occupational engagement and health outcomes among community-dwelling older adults. American Journal of Occupational Therapy, 66(3), 301-310.

- 15. Shirado, O., Shundo, M., Kaneda, K., & Strax, T. E. (1995). Outdoor Winter Activities of Spinal Cord-Injured Patients: With Special Reference to Outdoor Mobility. *American journal of physical* medicine & rehabilitation, 74(6), 408-414.
- 16. Morales, E., Gamache, S., & Edwards, G. (2014). Winter: Public Enemy# 1 for Accessibility EXPLORING NEW SOLUTIONS. Journal of Accessibility and Design for All, 4(1), 23.
- 17. Lemaire, E. D., O'Neill, P. A., Desrosiers, M. M., & Robertson, D. G. (2010). Wheelchair ramp navigation in snow and ice-grit conditions. Archives of physical medicine and rehabilitation, 91(10), 1516-1523.
- 18. Schneidert, M., Hurst, R., Miller, J., & Üstün, B. (2003). The role of environment in the International Classification of Functioning, Disability and Health (ICF). Disability & Rehabilitation, 25(11-12), 588-595.
- 19. Anaby, D., Lal, S., Huszczynski, J., Maich, J., Rogers, J., & Law, M. (2013). Interrupted Time Series Design: A Useful Approach for Studying Interventions Targeting Participation. *Physical &* occupational therapy in pediatrics.
- 20. Portney, L. G., & Watkins, M. P. (2008). Foundations of clinical research: applications to practice. Prentice Hall, Upper Saddle River.
- 21. Burke, W. J., Roccaforte, W. H., & Wengel, S. P. (1991). The short form of the Geriatric Depression Scale: a comparison with the 30-item form. J of geriatric psychiatry and neurology, 4(3), 173-178.
- 22. Nasreddine, Z. S., Phillips, N. A., Bédirian, V., Charbonneau, S., Whitehead, V., Collin, I., ... & Chertkow, H. (2005). The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. Journal of the American Geriatrics Society, 53(4), 695-699.
- 23. Law, M., Baptiste, S., Carswell, A., McColl, M. A., Polatajko, H., & Pollock, N. (2005). COPM Canadian Occupational Performance Measure. CAOT ACE: Ottawa, ON.
- 24. Baum, C. M., Edwards, D., & Michael, E. (2001). Activity card sort (ACS). Washington University School of Medicine.
- 25. Üstün, T. B., Chatterji, S., Kostanjsek, N., Rehm, J., Kennedy, C., Epping-Jordan, J., ... & Pull, C. (2010). Developing the World Health Organization disability assessment schedule 2.0. Bulletin of the World Health Organization, 88(11), 815-823.
- 26. Thorne, S. (2008). *Interpretive description* (Vol. 2). Left Coast Press.
- 27. Hsieh, H. F., & Shannon, S. E. (2005). Three approaches to qualitative content analysis. *Qualitative* health research, 15(9), 1277-1288.
- 28. Orellano, E., Colón, W. I., & Arbesman, M. (2012). Effect of occupation-and activity-based interventions on instrumental activities of daily living performance among community-dwelling older adults: A systematic review. American Journal of Occupational Therapy, 66(3), 292-300.